CLINICAL TRIAL: NCT01903447
Title: Negative Valence Brain Targets and Predictors of Anxiety and Depression Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, K. Luan Phan, MD, Professor of Psychiatry, Director, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-0325; R01MH101497 (NIH)
Record Dates: First submitted 2013-07-09; First posted 2013-07-19 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-01

CONDITIONS: Internalizing Psychopathologies (IPs) Depression and Anxiety
Keywords: Internalizing psychopathologies; Depression; Anxiety; MRI; medication treatment; psychotherapy; brain function
MeSH Terms: conditions — Ichthyosis prematurity syndrome; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SSRI (Active Comparator): sertraline: 100-200mg, citalopram 20-40mg, escitalopram 10-20mg, paroxetine 20-60mg; fluoxetine 20-80mg
  Interventions: Drug: SSRI
- CBT (Active Comparator): 12 weeks of individual cognitive behavioral therapy
  Interventions: Behavioral: CBT

INTERVENTIONS:
Drug: SSRI
  Arms: SSRI
Behavioral: CBT
  Arms: CBT

SUMMARY:
Internalizing psychopathologies (IPs) involving depression and anxiety are among the most prevalent, costly and disabling illnesses. Treatments for IPs are available but the extent to which individual patients respond is quite heterogeneous. Little information exists, particularly in the biological domain, which helps to explain individual differences in treatment response. IPs share similar patterns of dysfunction within the Fronto-Limbic Affect Regulation and Emotional Salience (FLARES) brain circuit, and two commonly used, 'gold standard' treatments - selective serotonin reuptake inhibitors (SSRIs) and cognitive behavioral therapies (CBTs) - are equally effective for both anxiety and depressive disorders, and appear to change brain activity in the same areas within the FLARES circuit. The overarching goal of the project is delineate what are common versus specific FLARE brain targets for SSRI and CBT and identify specific aspects of FLARE dysfunction that might better predict response to both and to a specific modality of treatment. This experiment integrates emotion and its interaction with cognition across several stages of emotional experience, encompassing studies that probe sensitivity to acute and potential threat and automatic and volitional forms of affect regulation in relation to the FLARES brain network.

We will enroll 200 patients presenting to our Mood and Anxiety Disorders Program seeking treatment for disabling 'anxiety, worry, depressed mood' (IPs, including those characterized as Not Otherwise Specified) and randomize them to a 12-week course of SSRI or CBT. Dimensional, transdiagnostic negative valence systems (NVS) constructs, including FLARES function, will be measured before and after each treatment. Specifically, the project will examine 2 Specific Aims: 1) Where and how do SSRI and CBT treatments exert their effects on NVS constructs?; and 2) Which NVS construct can predict the likelihood of success from SSRI and CBT treatment? Such findings can be used to guide the right patients to the right treatments with the highest likelihood of success. They also elucidate a pathophysiologically-driven mechanistic model of where and how treatments work in the brain and thus hasten the development of new treatments that target the underlying pathophysiology across internalizing conditions.

ELIGIBILITY:
Inclusion Criteria:

* Generally medically and neurologically healthy
* Chief complaint(s) of "anxiety, worry, and/or depressed mood

Exclusion Criteria:

* Current or past manic/hypomanic episode or psychotic symptoms
* Suicidal ideation
* Presence of contraindications (e.g., history of SSRI adverse events) or prior history of SSRI resistance (no response to > 2 SSRI trials with adequate duration and dose)
* Obsessive compulsive disorder (OCD)
* Current cognitive dysfunction (traumatic brain injury, mental retardation, dementia)
* Current alcohol and substance dependence
* Ongoing therapy/medication treatment of any kind outside of this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2013-12-13 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2018-02-21 (Actual)

PRIMARY OUTCOMES:
Brain NVS Construct Measure (Composite) | Change from Week 0 to Week 12
  Brain: functional magnetic resonance imaging (fMRI) BOLD percent signal change [PSC] within region of interests [ROIs: amygdala, bed nucleus of stria terminalis, striatum, hippocampus, anterior cingulate cortex (including dorsal, rostral, & subgenual subdivisions), anterior insula, ventro/dorso-medial prefrontal cortex, orbitofrontal cortex, ventro/dorso-lateral prefrontal cortex for Emotional Face Assessment Task (EFAT), Emotional Face Interference Task (EFIT), Contextual Threat Task (CTT), Emotion Regulation Task (ERT)

CONTACTS AND LOCATIONS:
Overall Officials: K. Luan Phan, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Kinney KL, Burkhouse KL, Chang F, MacNamara A, Klumpp H, Phan KL. Neural mechanisms and predictors of SSRI and CBT treatment of anxiety: A randomized trial focused on emotion and cognitive processing. J Anxiety Disord. 2021 Aug;82:102449. doi: 10.1016/j.janxdis.2021.102449. Epub 2021 Jul 10. PMID 34274600
- [Derived] Gorka SM, Young CB, Klumpp H, Kennedy AE, Francis J, Ajilore O, Langenecker SA, Shankman SA, Craske MG, Stein MB, Phan KL. Emotion-based brain mechanisms and predictors for SSRI and CBT treatment of anxiety and depression: a randomized trial. Neuropsychopharmacology. 2019 Aug;44(9):1639-1648. doi: 10.1038/s41386-019-0407-7. Epub 2019 May 6. PMID 31060042
- [Derived] Burkhouse KL, Gorka SM, Klumpp H, Kennedy AE, Karich S, Francis J, Ajilore O, Craske MG, Langenecker SA, Shankman SA, Hajcak G, Phan KL. Neural Responsiveness to Reward as an Index of Depressive Symptom Change Following Cognitive-Behavioral Therapy and SSRI Treatment. J Clin Psychiatry. 2018 Jun 12;79(4):17m11836. doi: 10.4088/JCP.17m11836. PMID 29894598